CLINICAL TRIAL: NCT04510207
Title: Multicenter, Randomized, Double Blind, Parallel Placebo Controlled, Phase III Clinical Trial to Evaluate the Protective Efficacy, Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccines (Vero Cell) in Healthy Population Aged 18 Years Old and Above
Brief Title: A Study to Evaluate The Efficacy, Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccines (Vero Cell) in Healthy Population Aged 18 Years Old and Above
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: G42 Healthcare company (Unknown); Abu Dhabi Health Services Company (Other Government); Wuhan Institute of Biological Products Co., Ltd (Industry); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CNBG2020003SQ
Record Dates: First submitted 2020-08-03; First posted 2020-08-12 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Investigational Vaccine 1 (Experimental): Participants will receive 2 doses of the inactivated SARS-CoV-2 vaccine (Vero cell) manufactured by WIBP according to the immunization schedule of D0 & D21.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell)
- Investigational Vaccine 2 (Experimental): Participants will receive 2 doses of the inactivated SARS-CoV-2 vaccine (Vero cell) manufactured by BIBP according to the immunization schedule of D0 & D21.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell)
- Placebo (Placebo Comparator): Participants will receive 2 doses of Placebo according to the immunization schedule of D0 & D21.
  Interventions: Biological: Placebo
- Investigational Vaccine 1b (Experimental): Participants will receive a booster dose of the inactivated SARS-CoV-2 vaccine (Vero cell) manufactured by WIBP after 3 months following two doses of immunization.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell)
- Investigational Vaccine 2b (Experimental): Participants will receive a booster dose of the inactivated SARS-CoV-2 vaccine (Vero cell) manufactured by BIBP after 3 months following two doses of immunization.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell)
- Placebo-b (Placebo Comparator): Participants will receive a booster dose of Placebo after 3 months following two doses of immunization.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) — The inactivated SARS-CoV-2 Vaccine (Vero cell) manufactured by WIBP
  Arms: Investigational Vaccine 1; Investigational Vaccine 1b
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) — The inactivated SARS-CoV-2 Vaccine (Vero cell) manufactured by BIBP
  Arms: Investigational Vaccine 2; Investigational Vaccine 2b
Biological: Placebo — The placebo of inactivated SARS-CoV-2 Vaccine (Vero cell) manufactured by WIBP
  Arms: Placebo; Placebo-b

SUMMARY:
This is a multicenter, randomized, double blind, parallel placebo controlled, phase 3 clinical trial to evaluate the protective efficacy, safety and immunogenicity of inactivated SARS-CoV-2 vaccines in healthy population 18 years old and above.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the protective efficacy, safety and immunogenicity of inactivated SARS-CoV-2 vaccines in healthy population 18 years old and above. The participants were randomized into three groups of investigational vaccine 1, investigational vaccine 2 and placebo in a 1:1:1 ratio.2 doses of the investigational vaccine or placebo are inoculated into the deltoid muscle of the either arm according to the vaccination schedule of D0 & D21 (+7 days).According to the immune durability results in Phase I/II study, and cross-neutralization assay results, a third dose (booster dose) generates a better immune response and is estimated to offer better protection, therefore, a booster dose will be given after 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 years old and above.
2. By asking for medical history and physical examination, the investigator judged that the health condition is well.
3. Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 3 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
4. During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan.
5. With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

1. Confirmed acute cases of SARS-CoV-2 Infection.
2. Have a history of SARS, MERS infection (self-report, on-site inquiry).
3. Positive urine pregnancy test result.
4. Fever (body temperature > 37.0 ℃), dry cough, fatigue, nasal obstruction, runny nose, pharyngeal pain, myalgia, diarrhea, shortness of breath and dyspnea occurred within 14 days before vaccination.
5. Axillary body temperature > 37.0 ℃ before vaccination.
6. Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS-CoV-2 vaccine have occurred.
7. Has a history of convulsion, epilepsy, encephalopathy or mental illness or family history.
8. With congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
9. With severe liver diseases, severe kidney diseases defined as eGFR less than 60, uncontrollable hypertension (systolic blood pressure >150 mmHg, diastolic blood pressure > 90 mmHg), diabetic complications, malignant tumors, various acute diseases, or acute attack period of chronic diseases.
10. Has been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases.
11. With known or suspected diseases include acute respiratory diseases (e.g. influenza like illness, acute cough, sore throat), severe cardiovascular diseases, liver and kidney diseases, and malignant tumors.
12. Has a history of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease).
13. Receiving anti-TB therapy.
14. Patients receiving immunotherapy or inhibitor therapy within 3 months (continuous oral or infusion for more than 14 days).
15. Live attenuated vaccine is inoculated within 1 month before this vaccination, other vaccines are inoculated within 14 days before this vaccination.
16. Received blood products within 3 months before this vaccination
17. Received other research drugs within 6 months before this vaccination.
18. Other circumstances judged by investigators that are not suitable for this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44101 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of COVID-19 cases after two-doses of vaccination | From14 days after the second dose to 6 month after the second dose
The incidence of COVID-19 cases after the booster dose of immunization | From 14 days after the booster dose

SECONDARY OUTCOMES:
The incidence of severe cases of COVID-19 and deaths accompanied by COVID-19 after two-doses of vaccination | From 14 day after the second dose to 6 month after the second dose
The incidence of severe cases of COVID-19 and deaths accompanied by COVID-19 after two-doses of vaccination | From 14 day after the booster dose
The incidence of any adverse reactions/events | 28 days after each immunization
The incidence of serious adverse events (SAE) | From the beginning of the first dose to 12 months after the second immunization
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 14 days after full course of immunization
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 14 days after full course of immunization
The Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody | 14 days after full course of immunization
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 28 days, 3rd month, 6th month, 9th month, and 12th month after 2 doses of immunization
The 4-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 28 days, 3rd month, 6th month, 9th month, and 12th month after 2 doses of immunization
The Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody | 28 days, 3rd month, 6th month, 9th month, and 12th month after 2 doses of immunization
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 14 days, 28 days and 6th month after the booster dose
The 4-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 14 days, 28 days and 6th month after the booster dose
The Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody | 14 days, 28 days and 6th month after the booster dose

OTHER OUTCOMES:
the anti-SARS-CoV-2 neutralizing antibody protective level against COVID-19 | 14 days after 2 doses of vaccination
The occurrence of ADE | From the beginning of the first dose to 12 months after the second immunization

CONTACTS AND LOCATIONS:
Overall Officials: Walid A Zaher, MD, MSc,PhD, Study Director — G42 Healthcare company
Locations (6):
- Bahrain International Exhibition & Convention Centre Affiliated to Salymynia Medical Complex S, Sanābis, Bahrain
- Egypt (2):
  - Katameya Medical Center, Cairo
  - Vacsera health Care facilities , MoH, Cairo
- Prince Hamza Hospital, Amman, Jordan
- United Arab Emirates (2):
  - Sheikh Khalifa Medical City, SEHA, Abu Dhabi
  - Al Qarain Primary Health Care Centre-MOHAP, Sharjah city

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Kaabi N, Yang Y, Eldin Hussein S, Yang T, Abdalla J, Wang H, Lou Z, Chinese Center For Disease Control And Prevention, Bakkour A, Arafat A, China National Biotec Group Company Limited, Jiang Z, Tian Y, National Engineering Technology Research Center For Combined Vaccines Wuhan Institute Of Biological Products Co Ltd, Beijing Institute Of Biological Products Company Limited, Xiao P, Zaher W, Eltantawy I, Wang C, Xu G, Zhang Y, Yang X. Efficacy and Safety of a Booster Vaccination with Two Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: Results of a Double-Blind, Randomized, Placebo-Controlled, Phase 3 Trial in Abu Dhabi. Vaccines (Basel). 2023 Jan 30;11(2):299. doi: 10.3390/vaccines11020299. PMID 36851177
- [Derived] Luan N, Li T, Wang Y, Cao H, Yin X, Lin K, Liu C. Th2-Oriented Immune Serum After SARS-CoV-2 Vaccination Does Not Enhance Infection In Vitro. Front Immunol. 2022 Apr 8;13:882856. doi: 10.3389/fimmu.2022.882856. eCollection 2022. PMID 35464483
- [Derived] Al Kaabi N, Zhang Y, Xia S, Yang Y, Al Qahtani MM, Abdulrazzaq N, Al Nusair M, Hassany M, Jawad JS, Abdalla J, Hussein SE, Al Mazrouei SK, Al Karam M, Li X, Yang X, Wang W, Lai B, Chen W, Huang S, Wang Q, Yang T, Liu Y, Ma R, Hussain ZM, Khan T, Saifuddin Fasihuddin M, You W, Xie Z, Zhao Y, Jiang Z, Zhao G, Zhang Y, Mahmoud S, ElTantawy I, Xiao P, Koshy A, Zaher WA, Wang H, Duan K, Pan A, Yang X. Effect of 2 Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):35-45. doi: 10.1001/jama.2021.8565. PMID 34037666